CLINICAL TRIAL: NCT05164328
Title: Prospective Athlete's Heart Study: Long-term Assessment of the Determinants of Cardiac Remodelling and Its Clinical Consequences in Endurance Athletes
Brief Title: Prospective Athlete's Heart Study
Acronym: Pro@Heart
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Baker Heart and Diabetes Institute (Other); Victor Chang Cardiac Research Institute (Unknown); University Hospital, Antwerp (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, dr. Guido Claessen, Chair, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: 57241
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Athlete Heart
Keywords: Athlete; Atrial fibrillation; Arrhythmias; Cardiac remodelling; Cardiomyopathy; Genetics
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes: 1. Males and females aged 14-23 years old
  2. Athletes competing in endurance sports at national or international level for at least 2 years. Sports include:
     1. Triathlon
     2. Cycling
     3. Distance running (≥ 1500 meters)
     4. Rowing
     5. Swimming
  Interventions: Other: No intervention
- Non-athletes: 1. Males and females aged 14-23 years old
  2. Non athletes engaged in < 3 hours per week of physical activity
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The Pro@Heart (Prospective Athlete's Heart) study is an international multicentre long-term prospective trial. The primary objective of the Pro@Heart study is to investigate the impact of training load (i.e. accurately evaluated in term of type, frequency, duration and intensity) and genotype on the variability of structural, functional and electrical exercise induced cardiac remodeling (EICR) in young competitive endurance athletes. The second objective is to determine how EICR, training load and genotype are associated with physical performance, health benefits and cardiac pathology (e.g. exercise-related cardiomyopathies and arrhythmias) during follow-up over several decades.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 14-23 years old
2. Athletes competing in endurance sports at national or international level for at least 2 years. Sports include:

   1. Triathlon
   2. Cycling
   3. Distance running (≥ 1500 meters)
   4. Rowing
   5. Swimming
3. Non athletes engaged in < 3 hours per week of physical activity

Exclusion Criteria:

1. Medical history of cardiovascular disease
2. Current smoker of past history of smoking
3. Diabetes mellitus

Ages: 14 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes aged 14 to 23 years recruited from elite endurance sports programs and organisations including Cycling Vlaanderen, Triatlon Vlaanderen, Belgian Cycling, Cycling Australia, Rowing Australia and Athletics Australia and from sports performance centres including Nottebohm Antwerpen, Bakala Academy Leuven and Adlon Hasselt. Volunteers recruited by means of 'word of mouth' and social media campaigns within elite endurance sporting circles. Non-athletes consist of age and gender matched university and college students recruited from Australian and Belgian universities in addition to social media campaigns.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2015-06-23 (Actual); Primary Completion 2035-06-23 (Estimated); Study Completion 2040-06-23 (Estimated)

PRIMARY OUTCOMES:
Genotype | Baseline
  Rare and common variants in cardiomyopathy associated genes
Training load | Baseline to 20 years
  Duration and intensity of training
Atrial fibrillation | Baseline to 20 years
Ventricular arrhythmias | Baseline to 20 years
  Ventricular ectopic beats, non-sustained and sustained ventricular tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Guido Claessen, Prof. Dr., Study Chair — UZ Leuven
Locations (4):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerp
  - Jessa Ziekenhuis Hasselt, Hasselt, Limburg
  - UZ Leuven, Leuven, Vlaams Brabants

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Bosscher R, Dausin C, Janssens K, Bogaert J, Elliott A, Ghekiere O, Van De Heyning CM, Sanders P, Kalman J, Fatkin D, Herbots L, Willems R, Heidbuchel H, La Gerche A, Claessen G; Pro@Heart Consortium. Rationale and design of the PROspective ATHletic Heart (Pro@Heart) study: long-term assessment of the determinants of cardiac remodelling and its clinical consequences in endurance athletes. BMJ Open Sport Exerc Med. 2022 Mar 18;8(1):e001309. doi: 10.1136/bmjsem-2022-001309. eCollection 2022. PMID 35368514
- See also: Study Website — https://www.proatheart.be/en/pro-heart-the-prospective-athletes-heart-study/